CLINICAL TRIAL: NCT05024500
Title: Clinical, Respiratory, Peripheral, Muscle and Functionality Outcomes of Adult ICU Inpatients and Rehabilitation-center Outpatients With COVID-19
Brief Title: Clinical and Functional Outcomes of Critically Ill Patients With COVID-19
Acronym: COVIDPTcare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other); Coordination for the Improvement of Higher Education Personnel (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Ciência e Tecnologia de Pernambuco (Other)
Responsible Party: Principal Investigator, Shirley Lima Campos, Associate Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVIDPTcare
Record Dates: First submitted 2020-12-18; First posted 2021-08-27 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: three groups of treatments (A, B and C) are given so that one group receives only A while another group receives only B and the third group receives only C. All volunteers will be randomized to one of the three groups of treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: trial participants, data collectors and outcome assessors or committees will remain blinded to the patient assigned group of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADRSNet protocol (Experimental): ARDSnet protocol is the current, standard of care for ARDS. Its used by setting PEEP and the fraction of inspired oxygen (FiO2) to achieve the oxygenation goal (SpO2 ≥ 93% - accepting the range of 90-96%)
  Interventions: Other: ARDSNet table
- Driving Pressure (DP) (Experimental): setting PEEP after performing a modified alveolar recruitment maneuver followed by a decremental PEEP titration electing the level correspondent to the lowest driving pressure.
  Interventions: Other: Driving Pressure
- Electrical Impedance Tomography (EIT) (Experimental): After performing a modified alveolar recruitment maneuver, the PEEP decremental titration guided by the EIT will be set at the level above the intersection of the curves representing relative alveolar overdistention and collapse.
  Interventions: Other: Electrical Impedance Tomography

INTERVENTIONS:
Other: ARDSNet table — The setting of the lowest PEEP level and FiO2 match stated by the table to achieve a goal oxygenation.
  Arms: ADRSNet protocol
Other: Driving Pressure — The setting of the lowest PEEP level by the lowest correspondent driving pressure, which is defined by the difference of plateau pressure, after a modified alveolar recruitment maneuver.
  Arms: Driving Pressure (DP)
Other: Electrical Impedance Tomography — The setting of the PEEP level above the intersection of the curves representing relative alveolar overdistention and collapse, after a modified alveolar recruitment maneuver.
  Arms: Electrical Impedance Tomography (EIT)

SUMMARY:
People affected by Severe Acute Respiratory Syndrome (SARS) by COVID-19 virus my require a long lasting invasive mechanical ventilation life support. To prevent damages to the lungs a number of protective lung ventilation measures are taken, one of them encounters the positive end expiratory pressure (PEEP) titration. Up to date, it is unclear the best method to titrate PEEP considering this unconventional syndrome compared to other etiologies. In addition to the long lasting advanced life support and bedridden condition, other factors may affect respiratory and peripheral muscle function of these patients. Therefore, the investigators intend to follow up these patients randomized to one of the three-arm experimental PEEP titration and after ICU discharge their status on clinical, laboratory and physical functions assessments.

DETAILED DESCRIPTION:
Introduction: Coronavirus Disease 2019 (COVID-19), caused by Severe Acute Respiratory Syndrome - Coronavirus-2 (SARS-CoV-2) requires mechanical ventilatory (MV) life support. In this scenario, lung protective strategies have been recommended for avoiding ventilator induced lung injuries mainly by inappropriate positive end expiratory pressure (PEEP) titration. However, the best method of PEEP titration for these patients remains unclear, since its clinical and morphofunctional phenotype may differ from the conventional acute respiratory distress syndrome (ARDS) phenotype resulted from other etiologies. In addition, these patients' condition of long lasting MV dependency and bed restriction may lead to deterioration of respiratory and peripheral muscles functions.

Objective: To compare the clinical and laboratory evolution and the respiratory and peripheral muscle functions in mechanically ventilated patients with COVID-19 submitted to PEEP titration by the following methods: ARDSNet protocol, driving pressure (DP) and electrical impedance tomography (EIT), as well as following them up after hospital discharge.

Methods: This is a controlled, randomized, double blind clinical trial with 90 mechanically ventilated patients to be randomized in one of the 3 PEEP titration- related groups: ARDSNet protocol, Driving Pressure-DP (electing PEEP level by the lowest DP) and by the EIT (PEEP selected will be the closest level above the intercept point of cumulated collapse and overdistension percentage curves). Clinical, laboratory, oxygenation, ventilation, respiratory and regional mechanics data, as well as peripheral muscle outcomes (strength and functionality) will be monitored from intubation to extubation in the supine and prone position. The outcomes of respiratory and peripheral muscles functionality will be monitored for six months after hospital discharge. All ethical principles will be respected with either written Free and Consent Term by the patient or relatives at the intensive care phase or at the post ICU discharge phase. Data will be registered for posterior analysis, which considers the difference between groups with p <0.05.

Expected results: Based on this study, it is expected to identify the Peep titration method associated to the greater beneficial and less deleterious effects in critically ill patients on MV. Also to address appropriate lung protective ventilation strategy for these patients and to detect respiratory and peripheral muscle disorders as early as possible in critically ill survivors.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated patients due to acute respiratory failure associated to COVID-19 confirmed or suspected cases

Exclusion Criteria:

* consent refusal by patient, family or doctor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-07-11 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Murray Score (LIS) | 4 hours
  Scoring system for lung injury including hypoxemia, respiratory system compliance, chest radiographic findings and level of PEEP. The minimum value is zero and the maximum value is sixteen. The higher the score the worse outcome.
Potential lung recruitment measured during electrical impedance tomography | 4 hours
  to quantify lung ventilation distribution

SECONDARY OUTCOMES:
Length of days in intensive care unit (ICU days) | Through study completion, an average of 1 year
  to quantify the number of days spent in a critical care unit
Work of breathing (WOB) measured during surface electromyography | 4 hours
  measured in root-mean-squared electromyography signals
Duration of mechanical ventilation (MV days) | Through study completion, an average of 1 year
  to quantity the number of days with use of invasive mechanical ventilation in inpatients.
ICU Mortality | Through study completion, an average of 1 year
  to quantify number of living days between ICU admission and deceased status
respiratory muscle strength | Through study completion, an average of 1 year
  maximal static respiratory mouth pressures
Forced vital capacity (FVC) measured during spirometry | Through study completion, an average of 1 year
  measures obtained by spirometry in outpatients
diaphragmatic mobility measured during ultrasonography | Through study completion, an average of 1 year
  diaphragmatic excursion expressed in millimeters
diaphragmatic thickening measured during ultrasonography | Through study completion, an average of 1 year
  diaphragmatic thickening expressed in millimeters
breathing pattern measured during airway flowmeter | Through study completion, an average of 1 year
  a device to quantify airway flow
peripheral muscle strength I | Through study completion, an average of 1 year
  to be evaluated by Medical Research Council's scale. The minimum score is 0 and the maximum is 60. The higher the score, the better outcome.
peripheral muscle strength II | Through study completion, an average of 1 year
  to be evaluated by a handgrip dynamometers in outpatients
peripheral muscle strength III | Through study completion, an average of 1 year
  to be evaluated by a handheld dynamometer in outpatients
six-minute walk test (6WT) | Through study completion, an average of 1 year
  sub-maximal exercise test used to assess aerobic capacity and endurance in outpatients
functional capacity (Perme scale) | Through study completion, an average of 1 year
  The minimum score is 0 and the maximum is 32. The higher the score, the better outcome.
daily activities performance | Through study completion, an average of 1 year
  to be evaluated by Barthel Index in outpatients
quality of life measured by Short Form Health survey 36 | Through study completion, an average of 1 year
  score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Lima Campos, PhD, Study Director — Universidade Federal de Pernambuco
Locations (4):
- Brazil (4):
  - Hospital das Clinicas - UFPE, Recife, Pernambuco
  - Physical Therapy Department, Universidade Federal de Pernambuco, Recife, Pernambuco
  - Hospital da Mulher do Recife, Recife, Pernambuco
  - Hospital Geral Otavio de Freitas, Recife, Pernambuco

IPD SHARING:
Plan to Share IPD: Yes
* participant characteristics (age, gender)
  * clinical measurements (blood pressure, heart rate)
  * medical history
  * clinical laboratory results
  * images (X-rays)
  * adverse events (hemodynamic and respiratory instability, interruptions)
  * details of randomisation and treatment received
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: end of trial
Access Criteria: individual participant data (IPD) access will be granted by the PI after request review for approval via email. It will be shared with researchers and general public of interest on the subject for descriptive analyses related to our sample medical and clinical characteristics. A committee of researchers will be in charge of discussing the request before approving the access.

REFERENCES:
- [Background] Adhikari SP, Meng S, Wu YJ, Mao YP, Ye RX, Wang QZ, Sun C, Sylvia S, Rozelle S, Raat H, Zhou H. Epidemiology, causes, clinical manifestation and diagnosis, prevention and control of coronavirus disease (COVID-19) during the early outbreak period: a scoping review. Infect Dis Poverty. 2020 Mar 17;9(1):29. doi: 10.1186/s40249-020-00646-x. PMID 32183901
- [Background] Adler A, Arnold JH, Bayford R, Borsic A, Brown B, Dixon P, Faes TJ, Frerichs I, Gagnon H, Garber Y, Grychtol B, Hahn G, Lionheart WR, Malik A, Patterson RP, Stocks J, Tizzard A, Weiler N, Wolf GK. GREIT: a unified approach to 2D linear EIT reconstruction of lung images. Physiol Meas. 2009 Jun;30(6):S35-55. doi: 10.1088/0967-3334/30/6/S03. Epub 2009 Jun 2. PMID 19491438
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Frerichs I, Becher T, Weiler N. Electrical impedance tomography imaging of the cardiopulmonary system. Curr Opin Crit Care. 2014 Jun;20(3):323-32. doi: 10.1097/MCC.0000000000000088. PMID 24739268
- [Background] Fumagalli J, Berra L. What does the Acute Respiratory Distress Syndrome trial (ART) teach us?-it is time for precision medicine and precision trials in critical care! J Thorac Dis. 2018 Mar;10(3):1300-1303. doi: 10.21037/jtd.2018.03.31. No abstract available. PMID 29707281
- [Background] Goh KJ, Choong MC, Cheong EH, Kalimuddin S, Duu Wen S, Phua GC, Chan KS, Haja Mohideen S. Rapid Progression to Acute Respiratory Distress Syndrome: Review of Current Understanding of Critical Illness from Coronavirus Disease 2019 (COVID-19) Infection. Ann Acad Med Singap. 2020 Mar 16;49(3):108-118. PMID 32200400
- [Background] Huh JW, Jung H, Choi HS, Hong SB, Lim CM, Koh Y. Efficacy of positive end-expiratory pressure titration after the alveolar recruitment manoeuvre in patients with acute respiratory distress syndrome. Crit Care. 2009;13(1):R22. doi: 10.1186/cc7725. Epub 2009 Feb 24. PMID 19239703
- [Background] Liu S, Tan L, Moller K, Frerichs I, Yu T, Liu L, Huang Y, Guo F, Xu J, Yang Y, Qiu H, Zhao Z. Identification of regional overdistension, recruitment and cyclic alveolar collapse with electrical impedance tomography in an experimental ARDS model. Crit Care. 2016 May 3;20(1):119. doi: 10.1186/s13054-016-1300-y. PMID 27142073
- [Background] Murray JF, Matthay MA, Luce JM, Flick MR. An expanded definition of the adult respiratory distress syndrome. Am Rev Respir Dis. 1988 Sep;138(3):720-3. doi: 10.1164/ajrccm/138.3.720. No abstract available. PMID 3202424
- [Background] Sahetya SK, Hager DN, Stephens RS, Needham DM, Brower RG. PEEP Titration to Minimize Driving Pressure in Subjects With ARDS: A Prospective Physiological Study. Respir Care. 2020 May;65(5):583-589. doi: 10.4187/respcare.07102. Epub 2019 Nov 26. PMID 31772068
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Zheng YY, Ma YT, Zhang JY, Xie X. COVID-19 and the cardiovascular system. Nat Rev Cardiol. 2020 May;17(5):259-260. doi: 10.1038/s41569-020-0360-5. PMID 32139904
- [Background] Silveira LTYD, Silva JMD, Tanaka C, Fu C. Decline in functional status after intensive care unit discharge is associated with ICU readmission: a prospective cohort study. Physiotherapy. 2019 Sep;105(3):321-327. doi: 10.1016/j.physio.2018.07.010. Epub 2018 Aug 2. PMID 30342701
- [Derived] Novaes APL, Campos SL, Leite WS, Morais CC, de Andrade AFD, Goncalves ACE, Moraes F, Brandao DC. Comparison Among Three PEEP Titration Methods Monitored by Electrical Impedance Tomography in COVID-19. Respir Care. 2023 Dec 28;69(1):106-109. doi: 10.4187/respcare.10627. No abstract available. PMID 37580123